CLINICAL TRIAL: NCT02256202
Title: Pilot Study of Quality Assurance in Interventional Pain Therapy in the Lumbal Spinal Column. Non-randomised, Evaluative, Multicentral Study Concerning the Applicability of a Tablet-PC.
Brief Title: Quality Assurance of Electronic Data Capturing (EDC) in Pain Treatment
Status: Completed | Type: Observational
Sponsor: Qualitouch-HC Foundation (Other)
Collaborators: Mundipharma Pte Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EDCINPT
Record Dates: First submitted 2014-09-25; First posted 2014-10-03 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Interview — Monitoring interviews to show medical and economic advantages of given therapy

SUMMARY:
There are actually no standardized quality assurance procedures included in pain treatment processes.

In this observational, feasibility study the use of tablet-Personal Computer (PC) is tested in pain therapy centres using the validated questionnaire "Activity Index". The acceptance of electronic data capturing is tested in patients and therapy teams (doctors and nurses).

DETAILED DESCRIPTION:
Regarding the demand for a duly documented efficacy of the therapy applied, a standardized procedure is imperative to show the medical and economic advantages of a given therapy. To obtain valid results, it is necessary to use a standardized process, monitored with a validated questionnaire.

In this multi-center study the Activity Index Questionnaire will be tested regarding its outcome quality regarding usability and patient acceptance. Each center collects data of 10 patients with injection pain therapy. Each patient is interviewed twice and after the 2nd interview each patient will fill out a feasibility questionnaire. During the whole study, the use and consumption of oral analgetic drugs are monitored in a diary. The statistical Analysis is done descriptive. Before entering the study, each patient has to give informed consent to participate. National Registration Guidelines for post market surveillance will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Willingness for therapeutic pain injection in lumbar spine

Exclusion Criteria:

* Cognitive impairment, technical Problems in interviewing patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Back pain patients
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of Tablet-PC in interviewing pain patients | 6-12 months
  The feasibility of the Tablet-PC in EDC will be assessed by standardized interviews (three times) of the study doctor, the study nurse and the patient.

SECONDARY OUTCOMES:
Problems in application of EDC in Tablet-PC | 12 months
  We measure the Problems of the Application of the EDC, e.g. Patient can't ush the button to answer the questions, e.g. some patients do not understand a question. The answers are usually given by Likert scales.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Theiler, Principal Investigator — Stadtspital Triemli Zurich, Department of Rheumatology
Locations (1):
- Stadtspital Triemli, Zurich, Canton of Zurich, Switzerland